CLINICAL TRIAL: NCT04849325
Title: A Prospective, Multi-Center, Randomized Trial Comparing the IBS Titan™ Sirolimus-Eluting Iron Bioresorbable Peripheral Scaffold System vs. Standard Balloon Angioplasty for Treatment of Below-the-Knee Arteries: GENIUS TRIAL
Brief Title: IBS Titan vs. PTA in Patients With Infrapopliteal Arterial Stenosis or Occlusive Disease
Acronym: GENIUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotyx Medical (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBS-Titan-01
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS Titan (Experimental)
  Interventions: Device: Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™)
- Percutaneous Transluminal Angioplasty (PTA) (Active Comparator)
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA) Device

INTERVENTIONS:
Device: Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™) — Subjects in this arm will be treated with IBS Titan™.
  Arms: IBS Titan
Device: Percutaneous Transluminal Angioplasty (PTA) Device — Subjects in this arm will be treated with PTA device.
  Arms: Percutaneous Transluminal Angioplasty (PTA)

SUMMARY:
A prospective, multi-center, randomized trial to assess the safety and effectiveness of Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™) in treating patients with infrapopliteal arterial stenosis or occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must between 18 and 85 years old, without gender limit.
2. Patients who can understand the purpose of the trial, voluntarily participate in and sign the informed consent form, and complete the 1-year follow-up.
3. Subject has lower extremity atherosclerotic occlusive disease with symptomatic Critical Limb Ischemia (CLI).
4. Rutherford Becker Clinical Category 3-5.
5. The target lesion is below the popliteal artery (including bifurcation).
6. The target lesion is located in the proximal 2/3 of native infrapopliteal vessels or tibiofibular trunk.
7. The target lesion stenosis is ≥70% or occlusion of no more than two infrapopliteal arteries (including the anterior and/or posterior tibial and/or peroneal artery and/or tibiofibular trunk).
8. The length of target lesion is ≤200mm, which could be covered by no more than two stents, with vessel diameter of 2.25-4.25 mm.

Exclusion Criteria:

1. Severe renal insufficiency, hepatic dysfunction (Cr>2 times of normal limit or renal dialysis, ALT or AST > 5 times of normal limit).
2. Surgery in target vessel before treatment.
3. Volume reduction surgery in target vessel before treatment.
4. Thrombosis in target vessel, or acute thrombosis requiring thrombolysis and thrombectomy.
5. Systematic coagulation disorder or hypercoagulability.
6. Lower extremity arteries surgery or thrombolytic therapy in the ipsilateral extremity in the past 6 weeks.
7. Stroke occurs within 3 months before surgery, or stroke occurs with severe hemiplegia aphasia sequelae more than 3 months before treatment.
8. Acute myocardial infarction or angina pectoris within 30 days before treatment.
9. In-stent restenosis.
10. Guide wire cannot pass target lesion.
11. Previously treated with drug eluting balloon within 1 year before treatment.
12. More than two infrapopliteal arteries needed treatment.
13. The inflow tract (including ipsilateral iliac artery, femoral artery, popliteal artery) has lumen stenosis >30% with or without intervention.
14. The inflow tract (including ipsilateral iliac artery, femoral artery, popliteal artery) has > 150 mm stenosis or occlusion before treatment.
15. Aneurysm of lower extremity artery.
16. Thromboangiitis obliterans (Buerger's disease).
17. Significant (≥ 50% stenosis) lesion in a distal outflow artery that would be perfused by the target vessel and that requires treatment at the time of the index procedure.
18. Patients known to be allergic to aspirin, heparin, Plavix, contrast agents, Sirolimus, poly lactic acid polymer, iron, zinc and their degradation product, and those who cannot tolerate postoperative dual anti-platelet therapy.
19. Patients who have a history of disease related to iron overload or iron disorder, such as hereditary hemochromatosis, etc.
20. Patients who are participating in another clinical trial that has not yet completed its primary endpoint.
21. Pregnant or those who plan pregnancy during the clinical investigation follow-up period.
22. Angiography suggests intraoperative thromboendarterectomy, percutaneous transluminal rotational atherectomy or laser therapy are needed.
23. Patients have life expectancy ≤ 1 year.
24. Patients who are not suitable for participating the trial judged by investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary Patency Rate | 180 days
  Defined as freedom from total occlusion of target lesion and clinically driven target lesion revascularization (CD-TLR) of target lesion, and freedom from major amputation.

SECONDARY OUTCOMES:
All-cause mortality | 30 days, 180 days, 365 days
Incidence of Clinically-driven Target Vessel Revascularization (CD-TLR) | 30 days, 180 days, 365 days
  CD-TLR is defined as any TLR of target lesions associated with Rutherford category exacerbation and/or increasing in the size of preexisting wounds and/or the occurrence of new wounds.
Incidence of major amputation | 30 days, 180 days, 365 days
  Unplanned amputation of the lower limb above the ankle on the target lesion side
Rate of Device Success | Immediately after the procedure
  Device success is defined on a per device basis, as the achievement of successful delivery, deployment of stent at the intended infrapopliteal target site(s) and successful withdrawal of the delivery catheter.
Rate of Participants with Technical Success | Immediately after the procedure
  Defined as restoration of blood flow in the target vessel and angiogram indicates the residual stenosis <50%.
Rate of Participants with Procedural Success | Immediately after the procedure
  Defined as the combination of technical success, device success, and absence of procedural complications.
Late Lumen Loss | 180 days
Incidence of Target lesion restenosis | 30 days, 180 days, 365 days
  Defined as a reduction in the luminal diameter >50% by angiography or CTA within the treated lesion plus the 5-mm segments proximal and distal to it or, as a peak systolic velocity ratio (PSVR) >2.4 by DUS.
  Note 1: Doppler ultrasound will be performed at 30 days and 365 days, DSA angiography will be performed 180 days.
  Note 2: If the patient presented with CD-TLR in advance, i.e. the patient reached the endpoint in advance, the restenosis before reintervention was assessed.
Change in ankle-brachial index (ABI) compared to baseline (before treatment) | 30 days, 180 days, 365 days
Change in Rutherford-Becker category compared to baseline (before treatment) | 30 days, 180 days, 365 days
  Categories and Clinical Description (higher scores mean a worse outcome):
  Category 0 = Asymptomatic, no hemodynamically significant occlusive disease, Category 1 = Mild claudication, Category 2 = Moderate claudication, Category 3 = Severe claudication, Category 4 = Ischemic rest pain, Category 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, Category 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable.
Wound healing rate of ulcer patients | 30 days, 180 days, 365 days

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - People's Liberation Army General Hospital, Beijing
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The First People's Hospital of Changzhou, Changzhou
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Second Hospital of Shanxi Medical University, Taiyuan
  - General Hospital of Tianjin Medical University, Tianjin
  - Tianjin 4th Centre Hospital, Tianjin
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided